CLINICAL TRIAL: NCT00598585
Title: Phase 4 Study of the Use of Sildenafil (Viagra) to Alter Fatigue, Functional Status and Impaired Cerebral Blood Flow in Patients With Chronic Fatigue Syndrome.
Brief Title: Use of Sildenafil (Viagra) to Alter Fatigue, Functional Status and Impaired Cerebral Blood Flow in Patients With CFS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Charles Drew University of Medicine and Science (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Theodore Friedman, Professor, Charles Drew University of Medicine and Science
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 02-04-378-07
Record Dates: First submitted 2005-08-31; First posted 2008-01-22 (Estimated); Results first posted 2017-06-27 (Actual); Last update posted 2017-06-27 (Actual); Status verified 2017-04

CONDITIONS: Chronic Fatigue Syndrome
MeSH Terms: conditions — Fatigue Syndrome, Chronic | interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- sidenafil (Experimental): sidenafil
  Interventions: Drug: Sildenafil (Viagra)
- placebo (Placebo Comparator): placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sildenafil (Viagra) — 25 mg tid of either Sildenafil(Viagra) for first week. 50 mg tid of either Sildenafil (Viagra) for second week. 100 mg tid of either Sildenafil (Viagra) 3rd,4th, 5th and 6th week of study participation.
  Arms: sidenafil
Drug: Placebo — Placebo pills 3X/day for 6 weeks
  Arms: placebo

SUMMARY:
Use of Viagra to Alter Symptoms in Patients with Chronic Fatigue Syndrome (CFS)

DETAILED DESCRIPTION:
Use of Sildenafil (Viagra) to Alter Fatigue, Functional Status and Impaired Cerebral Blood Flow in Patients with Chronic Fatigue Syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Patients meeting the CDC definition of CFS.
* All races, ethnicities, socio-economic status (SES), and gender
* Age greater than 18 (because of concerns about radioactivity, we and the Cedars-Sinai and Harbor-UCLA IRBs have decided not to enroll subjects below the age of 18).
* Age less than 50. Because of concern of sildenafil exacerbating coronary artery disease, we will only enroll patients younger than 50.
* Able to provide informed consent.
* Willingness to be off all medicines and supplements for 3 weeks prior to the study.
* Patients with psychiatric disorders (see below) will be included, if they could be off their medications, and if their psychiatric diagnosis clearly occurred after their fatigue symptoms began.
* Patients with concurrent fibromyalgia will be allowed to participate if the meet diagnostic criteria for CFS.

Exclusion Criteria:

* Disabilities that would prevent them from participating in the study.
* Current use of prescription medicines (starting at 3 weeks prior to the study) and supplements (starting at 1 weeks prior to the study) except acetaminophen or aspirin. This includes herbal supplements and vitamins.
* Existing medical illnesses, such as heart disease, hypertension, cancer, rheumatological diseases, endocrinopathies or hormone replacement therapy, seizure disorders, severe obesity (BMI > 32 kg/m2),
* Severe psychiatric disorders including bipolar disorder, schizophrenia, dementia and previous or current diagnosis of alcohol or substance abuse within the past year. Patients with depression of such severity as to warrant treatment with anti-depressants will be excluded.
* Current abuse of illicit drugs or heavy ethanol use.
* Pregnant women will be excluded because of radioactivity exposure from the SPECT scans.
* Abnormal EKG
* Abnormal CBC, blood chemistries, thyroid function tests, and HIV, ANA, RF and ESR tests.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2002-07; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ted C Friedman, M.D., Ph.D., Principal Investigator — Charles Drew University of Medicine and Science
Locations (1):
- Charles Drew University of Medicine and Science, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Clinical Trial Research site — http://www.centerwatch.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Sildenafil: 25 mg tid of Sildenafil(Viagra) for first week. 50 mg tid of Sildenafil (Viagra) for second week. 100 mg tid of Sildenafil (Viagra) for 3rd,4th, 5th and 6th week of study participation.
- Placebo: Placebo: Placebo
Period: Overall Study
Arm/Group | Sildenafil | Placebo
Started | 6 | 6
Completed | 5 | 6
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Sildenafil: Sildenafil(Viagra): 25 mg tid of Sildenafil(Viagra) for first week. 50 mg tid of Sildenafil (Viagra) for second week. 100 mg tid of Sildenafil (Viagra) for 3rd,4th, 5th and 6th week of study participation.
- Placebo: Placebo: Placebo tid for 6 weeks
- Total: Total of all reporting groups
Arm/Group | Sildenafil | Placebo | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 39 (6) | 38 (9) | 38 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 1 | 2 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 5 | 4 | 9
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 6 | 6 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Fatigue Impact Scale at 6 Weeks
Description: change in fatigue impact scale there are 42 questions. Each question can be answered from 0 (no problem) to 4 (extreme problem), so a higher score indicates more severe fatigue impact. minimum score=0, maximum score =148 values are calculated at baseline and 6 months and the score at 6 months compared to baseline months is calculated
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sildenafil | Placebo
Number analyzed (Participants) | 5 | 6
units on a scale | -32.6 (31.5) | -1.5 (12.2)
Statistical Analysis 1: Comparison: Sildenafil vs Placebo; Test type: Superiority — unpaired test, the threshold for statistical significance was p= 0.05; p < 0.05, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | Sildenafil | Placebo
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/6
Other Adverse Events (participants affected / at risk) | 1/5 | 0/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sildenafil (N=5) | Placebo (N=6)
dizziness (Cardiac disorders) | 1 (1) | 0 (0) — patient became dizzy after taking lasix

LIMITATIONS AND CAVEATS:
small number of subjects enrolled in trial

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No